CLINICAL TRIAL: NCT01348698
Title: Evaluation of Diagnostic and Prognostic Molecular Markers in Adrenal Neoplasm
Brief Title: Evaluation of Molecular Markers in Adrenal Tumors
Status: Terminated | Type: Observational
Why Stopped: Slow/insufficient accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Naris Nilubol, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110149; 11-C-0149
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Results first posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-10

CONDITIONS: Adrenal Gland Neoplasms
Keywords: Adrenal Cancer; Pheochromocytoma; Functioning Tumor; Nonfunctioning Tumor; Gene Expression; Adrenal Tumor
MeSH Terms: conditions — Adrenal Gland Neoplasms; Pheochromocytoma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adrenal Gland Neoplasm: To collect adrenal tumor tissue biopsy samples in order to study and evaluate new methods that may help identify cancerous or precancerous cells. Participants who have a large tumor or one that secretes hormones will have standard surgery to remove the tumor.
  Interventions: Procedure: Tumor tissue biopsy; Procedure: Surgery

INTERVENTIONS:
Procedure: Tumor tissue biopsy — Participants whose tumor does not secrete hormones will have a tumor biopsy to collect tissue for the study.
Procedure: Surgery — Participants who have a large tumor or one that secretes hormones will have standard surgery to remove the tumor. Tissue will be collected for study.

SUMMARY:
Background:

- Tumors of the adrenal gland are common. Most of them are not cancerous. However, there are no tests that can accurately tell which adrenal tumors are cancerous and which are not. The only way to tell is to remove the tumor with surgery and then examine it. Researchers have been using new methods to study samples of adrenal tissue. These methods may help identify whether the cells are or may become cancerous without an operation. This information will help doctors determine which tumors will need to be removed.

Objectives:

- To collect adrenal tumor tissue biopsy samples in order to study and evaluate new methods that may help identify cancerous or precancerous cells.

Eligibility:

- Individuals at least 18 years of age who have an adrenal tumor that may or may not be cancerous.

Design:

* Participants will be screened with a physical examination, medical history, blood and urine tests, and imaging studies.
* Participants will be examined to determine whether they have a specific type of adrenal tumor

(pheochromocytoma).

* Participants whose tumor does not secrete hormones will have a tumor biopsy to collect tissue for study.
* Participants who have a large tumor or one that secretes hormones will have standard surgery to remove the tumor. Tissue will be collected for study.
* Researchers will examine the collected tissue. They will try to determine whether the cells are cancerous or may become cancerous.
* Participants will be asked to return to the National Institutes of Health Clinical Center every year for about 5 years. During these visits they will have imaging studies, lab tests, and a physical examination.

DETAILED DESCRIPTION:
Background:

* Adrenal neoplasms are common and are incidentally discovered in 4-10% of abdominal imaging studies.
* The majority of adrenal incidentalomas are cortical adenoma.
* Many patients with nonfunctioning adrenal incidentalomas undergo adrenalectomy to exclude a cancer diagnosis.
* There are no reliable clinical, radiographic or laboratory studies that accurately distinguish between localized benign and malignant adrenal neoplasm.
* This protocol is designed to determine the feasibility and accuracy of using novel molecular markers of malignant adrenal neoplasm in fine needle aspiration (FNA) biopsy and surgically resected samples.

Objectives:

* Primary Objectives:

  * To evaluate the feasibility of molecular testing in adrenal neoplasm FNA biopsy samples.
  * To determine the accuracy of novel diagnostic molecular markers in clinical adrenal FNA biopsy and surgically resected samples.
* Secondary Objectives:

  * To analyze the gene expression level relative to disease-free survival and overall survival in patients with adrenocortical carcinoma

Eligibility:

* An individual with an adrenal neoplasm greater than 2cm in size
* Age greater than or equal to 18 years
* Adults must be able to understand and sign the informed consent document

Design:

* Prospective observational study.
* Demographic, clinical, laboratory and pathologic data will be collected for each patient participant. Data will be securely stored in a computerized database.
* Patients will have biochemical testing to determine if their adrenal neoplasm is functioning or nonfunctioning.
* After their initial on-study evaluation, patients who are found to have a nonfunctioning adrenal tumor with a low risk of malignancy will be re-screened every year for 5 years with non-invasive imaging studies.
* Treatment of patients with an adrenal neoplasm will be performed based on standard clinical practice.
* Projected accrual will be 50 patients per year for a total of 10 years. Thus, we anticipate accruing 500 patients on this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. An individual with a primary localized adrenal neoplasm greater than 2 cm in size
  2. Age greater than or equal to 18 years
  3. Adults must be able to understand and sign the informed consent document
  4. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance score of 0-2.
  5. Patients must have laboratory and physical examination parameters within acceptable limits by standard of practice guidelines prior to biopsy or surgery Note: patients with suspected but unconfirmed adrenal neoplasm may be enrolled.

EXCLUSION CRITERIA:

1. Biochemically proven Pheochromocytoma
2. Women who are pregnant because of the possible side effects of radiation from computed tomography (CT)-guided biopsies to the unborn child.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals at least 18 years of age who have an adrenal tumor that may or may not be cancerous. An individual with an adrenal neoplasm greater than 2cm in size.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2011-05-04 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naris Nilubol, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kloos RT, Gross MD, Francis IR, Korobkin M, Shapiro B. Incidentally discovered adrenal masses. Endocr Rev. 1995 Aug;16(4):460-84. doi: 10.1210/edrv-16-4-460. PMID 8521790
- [Background] NIH state-of-the-science statement on management of the clinically inapparent adrenal mass ("incidentaloma"). NIH Consens State Sci Statements. 2002 Feb 4-6;19(2):1-25. PMID 14768652
- [Result] Toniato A, Boschin I, Bernante P, Foletto M, Guolo AM, Pelizzo MR, Opocher G, Ballotta E, Mantero F. Factors influencing the rising rates of adrenal surgery: analysis of a 25-year experience. Surg Endosc. 2009 Mar;23(3):503-7. doi: 10.1007/s00464-008-0061-3. Epub 2008 Jul 15. PMID 18626702

RESULTS

PARTICIPANT FLOW:
Groups:
- Adrenal Gland Neoplasm: Adrenal neoplasms are common and are incidentally discovered in 4-10% of abdominal imaging studies. Most adrenal tumors are not cancerous. The majority of adrenal incidentalomas are cortical adenoma. Many patients with nonfunctioning adrenal incidentalomas undergo adrenalectomy to exclude a cancer diagnosis. There are no reliable clinical, radiographic or laboratory studies that accurately distinguish between localized benign and malignant adrenal neoplasm.
Period: Overall Study
Arm/Group | Adrenal Gland Neoplasm
Started | 74
Completed | 2
Not Completed | 72
Not completed — Does not meet lesion size criteria | 1
Not completed — Death | 3
Not completed — PI decision to close study | 68

BASELINE CHARACTERISTICS:
Arm/Group | Adrenal Gland Neoplasm
Number analyzed (Participants) | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.33 (12.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 17
  White | 47
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 74

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Molecular Testing in Adrenal Neoplasm Fine Needle Aspiration (FNA) Samples
Description: Feasibility of molecular testing in adrenal neoplasm fine needle aspiration (FNA) samples was determined by immunohistochemistry. Ribonucleic acid and deoxyribonucleic acid was extracted from fine needle aspiration and tumor tissue samples to differentiate between normal and abnormal tissue.
Time Frame: 5 years
Population: Because the study was terminated due to poor accrual and all fine needle aspiration (FNA) samples were benign, molecular testing cannot be performed in the absence of cancerous tumors. Molecular testing was not done in any samples collected.
Arm/Group | Adrenal Gland Neoplasm
Number analyzed (Participants) | 0

2. Primary Outcome: Determine the Accuracy of Novel Diagnostic Molecular Markers in Clinical Adrenal Fine Needle Aspiration (FNA) Biopsy and Surgically Resected Samples
Description: Tumor tissue obtained via FNA and surgical resection were to be analyzed for molecular markers to help determine if cells were cancerous or may become cancerous.
Time Frame: 5 years
Population: as for outcome 1
Arm/Group | Adrenal Gland Neoplasm
Number analyzed (Participants) | 0

3. Secondary Outcome: To Analyze the Gene Expression Level Relative to Disease-free Survival and Overall Survival in Patients With Adrenocortical Carcinoma
Description: Gene expression levels were to be analyzed relative to disease free and overall survival in patients with adrenocortical carcinoma.
Time Frame: 5 years
Population: as for outcome 1
Arm/Group | Adrenal Gland Neoplasm
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 6 years and 58 days
Measure: Count of Participants; unit: Participants
Arm/Group | Adrenal Gland Neoplasm
Number analyzed (Participants) | 74
Participants | 3

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 6 years and 58 days.
Arm/Group | Adrenal Gland Neoplasm
All-Cause Mortality (participants affected / at risk) | 3/74
Serious Adverse Events (participants affected / at risk) | 3/74
Other Adverse Events (participants affected / at risk) | 0/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adrenal Gland Neoplasm (N=74)
Death (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT01348698/Prot_SAP_ICF_000.pdf